CLINICAL TRIAL: NCT04037267
Title: Endoscopic Intraventricular Hematoma Evacuation Surgery Versus External Ventricular Drainage for the Treatment of Patients With Moderate to Severe Intraventricular Hemorrhage: a Multicenter, Randomized, Controlled Trial
Brief Title: Endoscopic Intraventricular Hematoma Evacuation Surgery Versus EVD for IVH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Professor, Nanjing PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019NZKY-014-01
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Intraventricular Hemorrhage, Endoscopic Intraventricular Evacuation Surgery, Extraventricular Drainage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Treatment (Experimental): Endoscopy was performed using a rigid endoscope. The hematoma was removed by a technique using irrigation and aspiration. The ventricular drainage catheter was placed on the surgical side. Six hours after surgery, we administered 20,000 U urokinase with 5 ml saline every 8 hours through the catheter and the catheter was closed for 1 hour to allow drug-clot interaction and then reopened to allow for gravitational drainage. Subsequent CT scans were done for any safety concern or every 24 hours. Administration of urokinase was stopped when the CT scans showed that the circulation of cerebrospinal fluid is unobstructed. When CT scans showed that the intracerebral hematoma was significantly reduced and the circulation of cerebrospinal fluid is unobstructed, the catheter could be clamped for 24 h. If there was no acute intracranial pressure increase, the catheter could then be removed.
  Interventions: Procedure: endoscopic intraventricular evacuation surgery
- EVD Treatment (Active Comparator): The surgeons used a soft catheter to puncture in depth of about 5 cm. The next step was to fix the drainage catheter. Postoperative CT was done immediately to confirm positioning of the soft catheter and stability of the hematoma. Six hours or more after catheter placement, we administered 20,000 U urokinase with 5 ml saline every 8 hours and the catheter was closed for 1 h to allow drug-clot interaction and then reopened to allow for gravitational drainage. Subsequent CT scans were done for any safety concern or every 24 hours. Administration of urokinase was stopped when the CT scans showed that the circulation of cerebrospinal fluid is unobstructed. When CT scans showed that the intracerebral hematoma was significantly reduced and the circulation of cerebrospinal fluid is unobstructed, the catheter could be clamped for 24 h. If there was no acute intracranial pressure increase, the catheter could then be removed.
  Interventions: Procedure: endoscopic intraventricular evacuation surgery

INTERVENTIONS:
Procedure: endoscopic intraventricular evacuation surgery — According to the discussion between the patient and the doctor, the patient signed the consent form and voluntarily enrolled and subsequently the patient was included in the endoscopic intraventricular evacuation surgery group.

SUMMARY:
Intraventricular hemorrhage (IVH) accounts for about 20% of intracerebral hemorrhage, but its mortality rate is as high as 50%-80%. External ventricular drainage (EVD) can rapidly reduce intracranial pressure, but clinical practice found that drainage catheters are often blocked by blood clots and long-term thrombolytic therapy is likely to cause secondary bleeding. The application of neuroendoscopy in IVH has attracted more and more attention in recent years. Studies have shown that the use of neuroendoscopy for IVH evacuation (with EVD) has advantages over EVD alone. However, the cases of most current research are small and all of them are retrospective studies, which means lacking prospective clinical studies to provide high-quality evidence. Based on this, we intend to conduct a randomized, controlled, multi-center clinical trial to compare the prognosis of patients who undergo endoscopic IVH evacuation surgery versus those who undergo external ventricular drainage for moderate to severe IVH.

DETAILED DESCRIPTION:
Spontaneous Intraventricular hemorrhage (IVH) is defined as bleeding into the cerebral ventricular system caused by spontaneous rupture of brain arteries, veins and capillaries instead of trauma. IVH accounts for about 20% of cerebral hemorrhage, but its mortality rate is as high as 50%-80%. According to the results of the STICH trial, the prognosis of patients with IVH is worse than that of patients without IVH (p<0.00001); if patients with IVH have hydrocephalus, the prognosis is the worst.

According to the edition of 2015 Chinese multidisciplinary experts' consensus for spontaneous cerebral hemorrhage diagnosis and treatment and 2015 AHA/ASA spontaneous cerebral hemorrhage diagnosis and treatment guidelines, for patients with small amount of IVH without obstructive hydrocephalus, conservative treatment or continuous lumbar drainage can be effective. For patients with large amount of IVH (hematoma occupying more than 50% of the lateral ventricle, secondary obstructive hydrocephalus or obviously increased intracranial pressure), the occupancy effect is dramatic and patients are prone to suffering from hydrocephalus and cerebral palsy, in which circumstances urgent evacuation of hematoma is required, but it is controversial whether it is beneficial for the patients and whether it can improve the prognosis of patients.

As the regular treatment for IVH, external ventricular drainage (EVD) can rapidly reduce intracranial pressure, but clinical practice found that drainage catheters are often blocked by blood clots, and long-term thrombolytic therapy is likely to cause secondary bleeding. Usually, the catheters need to be removed or replaced one week after placement as for the increasing risk of infection.

The application of endoscopy in IVH has attracted more and more attention. Studies have shown that the use of endoscopy for IVH evacuation (with EVD) has advantages over EVD alone. The incidence of postoperative hydrocephalus and the need for ventricular-peritoneal shunt surgery is lower. However, the cases of most current research are small and all of them are retrospective studies. There are no such clinical trials registered at home and abroad, and that is, there is a lack of prospective high-quality clinical studies to further demonstrate the effect of endoscopic treatment for IVH.

Based on this, we intend to conduct a randomized, controlled, multi-center clinical trial to compare the prognosis of patients who undergo endoscopic IVH evacuation surgery versus those who undergo external ventricular drainage for moderate to severe IVH.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ranging from 18 to 70 years old; 2. Imaging examination shows deep brain hemorrhage breaking into the ventricles or primary intraventricular hemorrhage, and the amount of bleeding is large, more than 50% of the lateral ventricle or complete ventricle cast; 3. Graeb score > 4 points; 4. Voluntary signing of informed consent;

Exclusion Criteria:

* 1. Patients with a history of chronic obstructive pulmonary disease, coronary heart disease, chronic kidney disease, blood disorders, cancer, systemic autoimmune disease, or long-term oral corticosteroids; 2. Imaging examination shows cerebellum and brain stem hemorrhage; 3. Detected cerebrovascular diseases in CTA/MRA/MRV/DSA examinations (choose 1 or 2 examinations); 4. Ultra-early (within 72 hours) or late enhanced MRI suggests the presence of brain tumors; 5. Coagulopathy or long-term oral anticoagulant;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 956 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Survival of patients at 12 months postoperatively | 12 months

SECONDARY OUTCOMES:
Modified Rankin score | preoperative, one month, three months, six months, twelve months
  Modified Rankin score
Proportion of patients who need ventricular-peritoneal shunt Incidence of postoperative hydrocephalus | 0-12 month
  Proportion of patients who need ventricular-peritoneal shunt Incidence of postoperative hydrocephalus
Incidence of postoperative intracranial infection | 0-12 month
  Incidence of postoperative intracranial infection
Hospital stay | 0-12 month
  Hospital stay
Hospitalization expenses | 0-12 month
  Hospitalization expenses

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhu J, Tang C, Cong Z, Yang J, Cai X, Liu Y, Ma C. Endoscopic intraventricular hematoma evacuation surgery versus external ventricular drainage for the treatment of patients with moderate to severe intraventricular hemorrhage: a multicenter, randomized, controlled trial. Trials. 2020 Jul 13;21(1):640. doi: 10.1186/s13063-020-04560-3. PMID 32660530